CLINICAL TRIAL: NCT05067465
Title: Screening to Validate and Identify Nutrition-related Biomarkers for Definded Food Groups (Dairy Products, Whole Grain, Processed Meat, Vegetarian Sausage Alternatives)
Brief Title: Nutritional Biomarker Screening for Defined Food Groups
Acronym: Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, PhD, University of Jena
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12_21
Record Dates: First submitted 2021-09-07; First posted 2021-10-05 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Healthy Lifestyle
Keywords: dairy products, whole grains, sausage, soy

STUDY DESIGN:
Intervention Model Description: Standardized diet over five days (n = 4x40) and test meal on day 6 with postprandial profiling (n = 4x12):
  Four groups characterized by defined intake of:
  1. Milk and dairy products
  2. Whole-grain products (rich in soluble fibers)
  3. Sausage and processed meat (pork)
  4. Meat-free sausage and meat alternatives (based on egg, soy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Milk and dairy products (Experimental): Standardized diet over five days (n = 40) - composed of cow milk, cheese, cream cheese, cream, valess milk schnitzel
  Test meal on day 6 (n = 12) - composed of milk, cheese, cream cheese, cream
  Interventions: Dietary Supplement: Selected food groups
- Whole-grain products (rich in soluble fibers) (Experimental): Standardized diet over five days (n = 40) - composed of oatmeal, oat bran, oat milk, whole wheat pasta, whole wheat bread, hummus
  Test meal on day 6 (n = 12) - composed of oatmeal, oat bran, oat milk
  Interventions: Dietary Supplement: Selected food groups
- Sausage and processed meat (pork) (Experimental): Standardized diet over five days (n = 40) - composed of Lyoner (pig), Viennese (pig), minced meat (pig)
  Test meal on day 6 (n = 12) - composed of Lyoner (pig), Viennese (pig)
  Interventions: Dietary Supplement: Selected food groups
- Meat-free sausage and meat alternatives (based on egg, pea, soy) (Experimental): Standardized diet over five days (n = 40) - composed of Mortadella (egg-based), Viennese (egg-based), vegan mince (soy-based)
  Test meal on day 6 (n = 12) - composed of Mortadella (egg-based), Viennese (egg-based)
  Interventions: Dietary Supplement: Selected food groups

INTERVENTIONS:
Dietary Supplement: Selected food groups — Food groups
  1. Milk and dairy products
  2. Whole-grain products (rich in soluble fibers)
  3. Sausage and processed meat (pork)
  4. Meat-free sausage and meat alternatives (based on egg, soy)

SUMMARY:
The Biomarker study will be conducted (i) to establish biomarker profiles that reflect the daily diet and regularly dietary habits, (ii) to complement self-reported dietary habits and (iii) to reduce gaps between self-reported information and real dietary intake. The study aims to assess relationships between defined nutrient intake (four groups: 1. Milk and dairy products, 2. Whole-grain products (rich in soluble fibers), 3. Sausage and processed meat (pork), 4. Meat-free sausage and meat alternatives (based on egg, soy) and resulting biochemical markers in human samples (plasma, serum, 24 h urine). In a next step, we will focus on unraveling the connection of the established diet-related metabolites with biomarkers of health and disease status, with focus on cardiovascular diseases (CVD).

DETAILED DESCRIPTION:
Within the scope of the present study, biomarkers or biomarker profiles are to be identified which reflect the daily diet and eating habits (focus: mixed diet / Western diet, vegetarians, vegans) in order to supplement or complete the information from diet protocols.

The chosen study design enables relationships between a defined nutrient intake in the form of a standardized diet over five days (four groups with 40 subjects each; group 1: Milk and dairy products, group 2: Whole grain products (rich in soluble fiber), group 3: Sausage and processed meat (pork), group 4: Meat-free sausage and meat alternatives (based on egg, soy) and the resulting biochemical markers in the human samples (plasma, serum, whole blood, 24-hour urine).

In addition, one subgroup (n = 12) consumed a test meal with the study foods on day 6 after the 5-day standardized diet. Before the test meal (time 0) and at intervals of 30, 60, 120, 180 min, blood samples are taken (postprandial profiling) in order to examine the brief increase in nutrients from the study foods in the human samples.

The aim of the study is i) to validate already established biomarkers and ii) to identify new biomarkers / patterns.

In the further course of the study, the identified and validated nutrition-associated biomarkers are to be linked to parameters of the health and disease status, whereby in particular the connection to cardiovascular risk factors and endpoints is considered.

Furthermore, the study design enables an assessment of the physiological effects as a result of an increased intake of the selected food (groups).

ELIGIBILITY:
Inclusion Criteria:

* Females (before menopause) and males
* Age: 20 < 40 years
* BMI ≥ 18 < 25 kg/m2
* Participants must be subjectively healthy
* Compatibility to one of the four planned groups as confirmed by lifestyle and nutrition-related questionnaires plus food frequency protocol (FFP) over five days
* Precondition: stable eating habits at least one year before enrollment

Exclusion Criteria:

* Subjects with any acute or chronic disease (tumor, infection, other), gastrointestinal diseases, dia-betes mellitus (type I, II), chronic renal disease, diseases of the parathyroid, diseases necessitating regular phlebotomies
* Intake of additional dietary supplements (e.g. fish oil capsules, vitamins, minerals etc.)
* Weight loss or weight gain (> 3 kg) during the last three months before study begin
* Pregnancy or lactation
* Transfusion of blood in the last three months before blood sample taking

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Fatty acids, concentration in %fatty acid methyl esters | Change from baseline after 5 days of the standardised diet
  Fatty acids distribution in plasma lipids, inclusive odd-chain fatty acids

SECONDARY OUTCOMES:
1-methylhistidineanserine, concentration | Change from baseline after 5 days of the standardised diet
  Marker for meat consumption
3-methylhistidineanserine, concentration | Change from baseline after 5 days of the standardised diet
  Marker for meat consumption
Asymmetric dimethylarginine, concentration | Change from baseline after 5 days of the standardised diet
  Marker for meat consumption
Homoarginine, concentration | Change from baseline after 5 days of the standardised diet
  Marker for meat consumption
Trimethylamine N-oxide, concentration | Change from baseline after 5 days of the standardised diet
  Marker for meat consumption
Syringol sulfate, concentration | Change from baseline after 5 days of the standardised diet
  Biomarkers for smoked meat intake
Alkylresorcinol, concentration | Change from baseline after 5 days of the standardised diet
  Markers for consumption of whole grains
Wheat germ agglutinin, concentration | Change from baseline after 5 days of the standardised diet
  Marker for consumption of whole grains
Galactitol, concentration | Change from baseline after 5 days of the standardised diet
  Markers for consumption of dairy products
Galactonate, concentration | Change from baseline after 5 days of the standardised diet
  Markers for consumption of dairy products
Galactono-1,5-lactone, concentration | Change from baseline after 5 days of the standardised diet
  Markers for consumption of dairy products
3-phenyllactic acid, concentration | Change from baseline after 5 days of the standardised diet
  Markers for consumption of dairy products

OTHER OUTCOMES:
Body mass index, kg/m2 | Change from baseline after 5 days of the standardised diet
  Anthropometric data
Systolic blood pressure, mm Hg | Change from baseline after 5 days of the standardised diet
  Cardiovascular risk factor
Diastolic blood pressure, mm Hg | Change from baseline after 5 days of the standardised diet
  Cardiovascular risk factor
Total cholesterol, mmol/l | Change from baseline after 5 days of the standardised diet
  Cardiovascular risk factors
LDL cholesterol, mmol/l | Change from baseline after 5 days of the standardised diet
  Cardiovascular risk factors
HDL cholesterol, mmol/l | Change from baseline after 5 days of the standardised diet
  Cardiovascular risk factors
Triacylglcerides, mmol/l | Change from baseline after 5 days of the standardised diet
  Cardiovascular risk factors
High sensitive c-reactive protein, mg/l | Change from baseline after 5 days of the standardised diet
  Inflammation marker
Fasting glucose, mmol/l | Change from baseline after 5 days of the standardised diet
  Diabetes risk factor
Fasting insulin, mU/l | Change from baseline after 5 days of the standardised diet
  Diabetes risk factor

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dawczynski, PhD, Principal Investigator — Friedrich-Schiller-University Jena
Locations (1):
- Institute of Nutritional Sciences, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the study center — https://www.nuco.uni-jena.de/studien